CLINICAL TRIAL: NCT07320144
Title: Investigation of the Effects of a Biopsychosocial Approach Added to Physiotherapy on Stress, Sleep Disturbance, and Bruxism in Individuals With Temporomandibular Disorders
Brief Title: Effects of a Biopsychosocial Approach Added to Physiotherapy in Temporomandibular Disorders
Acronym: TMD-BPS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Betül Özata (Other)
Responsible Party: Sponsor-Investigator, Betül Özata, Physiotherapist, MSc Student, Istinye University
Organization: Istinye University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMD-BPS-2025; 2025310 (Other Grant/Funding Number: Istinye University Ethics Committee)
Record Dates: First submitted 2025-12-22; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Temporomandibular Disorders (TMD)
Keywords: Temporomandibular joint; Pain education; Bruxism; Sleep quality; Biopsychosocial approach
MeSH Terms: conditions — Temporomandibular Joint Disorders; Bruxism; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either physiotherapy alone or physiotherapy combined with a biopsychosocial approach.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physiotherapy (Active Comparator): Participants in this arm will receive a standardized physiotherapy program for temporomandibular disorders, including therapeutic exercises and manual therapy targeting the temporomandibular joint and associated musculoskeletal structures.
  Interventions: Other: Physiotherapy Program
- Physiotherapy Plus Biopsychosocial Approach (Experimental): Participants in this arm will receive the same physiotherapy program combined with a biopsychosocial intervention including pain education, stress management strategies, and sleep hygiene education.
  Interventions: Other: Physiotherapy Program; Other: Biopsychosocial Intervention

INTERVENTIONS:
Other: Physiotherapy Program — A standardized physiotherapy program including therapeutic exercises and manual therapy targeting the temporomandibular joint and related musculoskeletal structures.
Other: Biopsychosocial Intervention — A biopsychosocial intervention including pain neuroscience education, stress management strategies, and sleep hygiene education.
  Arms: Physiotherapy Plus Biopsychosocial Approach

SUMMARY:
Temporomandibular disorders are conditions that affect the jaw joint and surrounding muscles and may cause pain, limited jaw movement, stress, sleep problems, and teeth grinding. Physiotherapy is commonly used to manage these problems, but psychological and social factors may also influence symptoms.

The purpose of this study is to examine whether adding a biopsychosocial approach to physiotherapy improves stress levels, sleep quality, and bruxism in individuals with temporomandibular disorders. Participants will receive either physiotherapy alone or physiotherapy combined with education about pain, stress management, and sleep habits. The results of this study may help improve treatment strategies for people with temporomandibular disorders.

DETAILED DESCRIPTION:
This randomized interventional study aims to investigate the effects of adding a biopsychosocial approach to physiotherapy in individuals with temporomandibular disorders. Temporomandibular disorders are multifactorial conditions influenced by physical, psychological, and social factors. While physiotherapy is effective in reducing pain and improving function, psychosocial factors such as stress, sleep disturbance, and bruxism may contribute to symptom persistence.

Participants will be randomly assigned to one of two groups. The control group will receive a standardized physiotherapy program including therapeutic exercises and manual therapy targeting the temporomandibular joint and related musculoskeletal structures. The intervention group will receive the same physiotherapy program in addition to a biopsychosocial intervention consisting of pain neuroscience education, stress management strategies, and sleep hygiene education.

Outcome measures will include stress levels, sleep disturbance, and bruxism severity as primary outcomes, and pain intensity and jaw function as secondary outcomes. Assessments will be conducted at baseline and after the intervention period. This study is expected to provide evidence on the effectiveness of integrating a biopsychosocial approach into physiotherapy for temporomandibular disorders.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with temporomandibular disorders
* Age between 18 and 65 years
* Presence of stress, sleep disturbance, or bruxism symptoms
* Ability to understand and follow study instructions
* Willingness to participate and provide informed consent

Exclusion Criteria:

* History of temporomandibular joint surgery
* Presence of neurological, rheumatological, or systemic diseases affecting the musculoskeletal system
* Current orthodontic treatment
* Use of medications that may affect pain perception or sleep
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Stress Level | Baseline and 6 weeks
  Stress level will be assessed using a validated self-reported questionnaire to evaluate perceived stress in individuals with temporomandibular disorders.

SECONDARY OUTCOMES:
Sleep Disturbance | Baseline and 6 weeks
  Sleep disturbance will be assessed using a validated questionnaire evaluating sleep quality and sleep-related problems.
Bruxism Severity | Baseline and 6 weeks
  Bruxism severity will be evaluated based on self-reported measures assessing teeth grinding and clenching behaviors.

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the study involves sensitive personal and health-related information, and data sharing was not included in the original ethical approval. Data will be used solely for the purposes of this study and related scientific publications.